CLINICAL TRIAL: NCT04030520
Title: Improving Uptake and Adherence to HIV Prevention Services With PrEP, HIV Self- Testing and Adherence Support for Very High Risk HIV-negative Young Women Aged 15-24 in Kampala, Uganda
Brief Title: Improving Uptake and Adherence to HIV Prevention Services With Pre-exposure Prophylaxis (PrEP), HIV Self- Testing and Adherence Support for Very High Risk HIV-negative Young Women Aged 15-24 in Kampala, Uganda
Acronym: POPPi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: MRC/UVRI and LSHTM Uganda Research Unit (Other); Medical Research Council (Other Government); London School of Hygiene and Tropical Medicine (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MH114523; R34MH114523 (NIH)
Record Dates: First submitted 2019-07-08; First posted 2019-07-24 (Actual); Results first posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): participants will receive a behavioral intervention including counseling and offer of HIV oral fluid self test and PrEP
  Interventions: Behavioral: POPPi
- comparison (Active Comparator): participants will be not be offered HIV oral fluid self test but receive counseling, condoms and offered PrEP
  Interventions: Behavioral: Comparison

INTERVENTIONS:
Behavioral: POPPi — behavioral intervention with offer of HIV self test
  Arms: intervention
Behavioral: Comparison — standard of care
  Arms: comparison

SUMMARY:
The main aim is to develop and assess an intervention to enhance initiation and adherence to PrEP among HIV negative young women of high risk (YWHR). The specific aims are (1) To conduct formative research to enhance our understanding of the dynamics of the social and sexual networks, and context of young HIV-uninfected women (aged 15-24) engaged in high risk sexual behavior in Kampala, Uganda (2) Document barriers and opportunities for PrEP uptake and adherence as well as repeat HIV testing by self test; (3) To develop and test a socially and culturally acceptable and feasible prevention intervention on uptake and adherence to PrEP and HIV self-testing for young women at high risk for HIV.

ELIGIBILITY:
Inclusion Criteria:

* Female age 15- to 24-years old
* Engaging in high-risk sexual behavior having had sex at least once in last three months, --HlV-negative
* Agree to participate in a minimum of four interviews over a 12-month period; including baseline
* Willing to receive services at Good Health for Women Project (GHWP)
* For those initiating PrEP (Truvada):
* Participants should have immunity to Hepatitis B infection and serum creatinine before
* Contra-indications for starting Truvada to be considered include Creatinine > 1.2 ( (mgldl) or 0.106 (mmolil) and a weight below 35kg.

Exclusion Criteria:

* Inability to consent to participation in the study
* Condition impeding participation in the study, including severe mental reason to the discretion of the principal investigator, cognitive impairment or illness; serious medical illness or developmental disability and any other reason to the discretion of the principal investigator.

Ages: 15 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2021-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel King, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Uganda Virus Research Institute, Entebbe, Uganda

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: participants will receive a behavioral intervention including counseling and offer of HIV oral fluid self test and PrEP
  POPPi behavioral intervention: behavioral intervention with offer of HIV self test
- Comparison: participants will be not be offered HIV oral fluid self test but receive counseling, condoms and offered PrEP
  POPPi behavioral intervention: behavioral intervention
Period: Overall Study
Arm/Group | Intervention | Comparison
Started | 30 | 30
Completed | 30 (we completed the target number) | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intervention: participants received a behavioral intervention including counseling and offer of HIV oral fluid self test and PrEP POPPi behavioral intervention: behavioral intervention with offer of HIV self test
- Comparison: participants were not be offered HIV oral fluid self test but receive counseling, condoms and offered PrEP POPPi behavioral intervention: behavioral intervention
- Total: Total of all reporting groups
Arm/Group | Intervention | Comparison | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14 | 14 | 28
  Between 18 and 65 years | 16 | 16 | 32
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.5 (2.1) | 19.5 (2.3) | 19.5 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ugandan | 30 | 30 | 60
Region of Enrollment [Number; unit: participants]
  Uganda | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Initiation of PrEP
Description: Initiation of PrEP using the pharmacy records indicating PrEP received by participants.
Time Frame: 6 months
Population: Number of participants who initiated PrEP using pharmacy pill count records.
Measure: Count of Participants; unit: Participants
Groups:
- Intervention; Comparison: number of participants initiating PrEP
Arm/Group | Intervention | Comparison
Number analyzed (Participants) | 30 | 30
Participants | 18 | 21

2. Primary Outcome: Adherence to PrEP
Description: Adherence to PrEP using hair analysis measured by the concentration of antiretroviral drug in strands of hair. The results will be measured per participant using concentration in nanograms/milligrams. The number of participants who showed a positive drug concentration in nanograms/milligrams is reported.
Time Frame: 12 months
Population: This is the number of participants who took PrEP and had samples tested at endline (12 months)
Measure: Count of Participants; unit: Participants
Groups:
- Intervention; Comparison: Uptake of PrEP
Arm/Group | Intervention | Comparison
Number analyzed (Participants) | 20 | 20
Participants | 19 | 18

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- Intervention: behavioral intervention
Arm/Group | Intervention | Comparison
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-12): https://cdn.clinicaltrials.gov/large-docs/20/NCT04030520/Prot_SAP_000.pdf